CLINICAL TRIAL: NCT05323630
Title: Evaluation of the Use of the Renuvion APR System in the Labia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apyx Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APX-22-02
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Labia Enlarged; Labium; Hypertrophy
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, single arm, evaluator-blinded study of the subjects undergoing a procedure with the Renuvion APR System in the labia. Follow-up visits will occur 1D Contact, 14D, 30D, 90D, and 180D post-procedure. Images will be captured at baseline and all follow-up visits.
  Three experienced, independent blinded photographic reviewers will perform a qualitative analysis/review of pre-treatment and post-treatment sets of images for each subject. Images will be provided in a blinded and randomized order. Each blinded reviewer will choose which is the before image and which is the after. Success will be correct identification of before and after by at least 2 of the 3 reviewers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Procedure with the Renuvion APR System in the labia (Other): The labia procedure utilizing the Renuvion APR system will be performed per the investigator's standard clinical practice.
  Interventions: Device: Renuvion APR System

INTERVENTIONS:
Device: Renuvion APR System — The Apyx Medical Corporation Renuvion/J-Plasma helium plasma family of products has received FDA clearance under 510(k) numbers K191542, K192867 for the cutting, coagulation, and ablation of soft tissue.

SUMMARY:
Labiaplasty is a procedure aimed at reducing lax or loose skin in the labia majora and/or minora due to childbirth, trauma, aging, genetics, or congenital disease.

DETAILED DESCRIPTION:
While traditional surgical procedures have been associated with complications such as dehiscence, hematoma, flap necrosis, narrowed introitus, and pain and asymmetry, correction with RF energy has shown minimal complication rates with high patient satisfaction. This study aims to evaluate the use of the Renuvion APR System for use as a minimally invasive alternative to surgical labiaplasty.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects, ages 35 - 70 years old.
* ASA Physical Status Classification System Class I and Class II subjects.
* Labial protrusion Class II and Class III (MOTAKEF scale)12.
* Females who do not desire traditional invasive surgery.
* Understands and accepts the obligation not to undergo any other procedures or treatments in the areas to be treated during study participation.
* Absence of physical conditions unacceptable to the investigator.
* Females of childbearing potential who are sexually active must be willing to use an approved method of birth control during study participation.
* Willing and able to comply with protocol requirements, including study-required images/photos, assessments/measurements, and returning for follow-up visits.
* Willing to release rights for the use of study photos, including in publication.
* Able to read, understand, sign, and date the informed consent.

Exclusion Criteria:

* Labial protrusion Class I (MOTAKEF scale).
* Subjects presenting with ASA Physical Status Classification System Classes III or higher.
* Pregnant, lactating, or plans to become pregnant during study participation.
* Known hypersensitivity or allergy to tumescent anesthetic (lidocaine/ epinephrine).
* Previous treatment in the study treatment area.
* Active systemic or local skin disease that may alter wound healing.
* Significant or uncontrolled medical condition that in the opinion of the investigator participation in the study may compromise the patient's health.
* Known susceptibility to keloid formation or hypertrophic scarring.
* Cancerous or pre-cancerous lesions in the area to be treated.
* Possesses a surgically implanted electronic device (i.e., pacemaker).
* Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in the past two years.
* Participation in any other investigational study within 30 days prior to consent and throughout study participation.
* Subject who, in the opinion of the investigator, is not an appropriate candidate for the study.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul G Ruff, MD, Principal Investigator — West End Plastic Surgery
Locations (1):
- Allison Plastic Martinez, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were no pre-assignments, but 7 subjects were treated with the APR-15-TP Handpiece and 3 of the subjects were treated with the Micro Handpiece launched after the study began.
Groups:
- Procedure With the Renuvion APR System in the Labia (APR-15-TP): The labia procedure utilizing the Renuvion APR system will be performed per the investigator's standard clinical practice. The APR-15-TP Handpiece was used in this group.
  Renuvion APR System: The Apyx Medical Corporation Renuvion/J-Plasma helium plasma family of products has received FDA clearance under 510(k) numbers K191542, K192867 for the cutting, coagulation, and ablation of soft tissue.
- Procedure With the Renuvion APR System in the Labia (Micro): The labia procedure utilizing the Renuvion APR system will be performed per the investigator's standard clinical practice. The Micro Handpiece was used in this group.
  Renuvion APR System: The Apyx Medical Corporation Renuvion/J-Plasma helium plasma family of products has received FDA clearance under 510(k) numbers K191542, K192867 for the cutting, coagulation, and ablation of soft tissue.
Period: Overall Study
Arm/Group | Procedure With the Renuvion APR System in the Labia (APR-15-TP) | Procedure With the Renuvion APR System in the Labia (Micro)
Started | 7 | 3
Completed | 7 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Procedure With the Renuvion Micro System in the Labia: The labia procedure utilizing the Renuvion Micro system will be performed per the investigator's standard clinical practice.
- Total: Total of all reporting groups
Arm/Group | Procedure With the Renuvion APR System in the Labia | Procedure With the Renuvion Micro System in the Labia | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 3 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: Years] | 41 (4) | 41 (8.5) | 41 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 3 | 1 | 4
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 3 | 10
BMI [Mean (Full Range); unit: kg/m2] | 25.246 [19.63 to 31.16] | 26.773 [25.13 to 27.72] | 25.704 [19.63 to 31.16]

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Change Between Baseline and Follow-up Images as Determined by a Masked, Qualitative Assessment of Photographs at 90-days and 180-days Post-treatment Compared to Baseline.
Description: Three experienced, blinded photographic reviewers performed a qualitative analysis/review of pre-treatment and post-treatment sets of images at 90-days and 180-days post-treatment compared to baseline for each subject. Images were provided in a blinded and randomized order. Each blinded reviewer choose which set of images were the post-treated Renuvion images of the labia. Change was assessed as success with success being the correct identification of treated labia images by at least 2 of the 3 reviewers.
Time Frame: Day 90, Day 180
Measure: Count of Units; unit: Sets of B/A Images analyzed
Units Other Than Participants: Sets of B/A Images analyzed
Arm/Group | Procedure with the Renuvion APR System in the labia (APR-15-TP) | Procedure with the Renuvion APR System in the labia (Micro)
Number analyzed (Participants) | 7 | 3
Number analyzed (Sets of B/A Images analyzed) | 14 | 6
Sets of B/A Images analyzed | 4 | 4

2. Secondary Outcome: Analysis of Morphometric Labia Measurements at D180.
Description: Analysis by anatomical measurements of the labia majora and minora at D180.
Time Frame: Day 180
Measure: Median (Standard Deviation); unit: cm
Arm/Group | Procedure with the Renuvion APR System in the labia (APR-15-TP) | Procedure with the Renuvion APR System in the labia (Micro)
Number analyzed (Participants) | 7 | 3
cm
  Sulcus Length of Labia Majora (Posterior to Anterior Margins) Day 180 | 10.0 (0.6) | 10.5 (0.7)
  Introital Opening to Most Anterior Projecting Edge of the Labia Minora Day 180 | 1.3 (0.6) | 1.3 (0.8)
  Posterior Border of the Sulcus to the Fornix Day 180 | 0.9 (0.2) | 0.9 (0.1)
  Inter-Labial Sulcus Length Day 180 | 9.0 (1.0) | 7.6 (1.5)
  Resting Projection of Labia Minora Beyond Labia Majora Day 180 | 0.7 (0.5) | 0.8 (0.5)
  Maximum Projection of the Labia Minora Day 180 | 1.8 (0.8) | 1.8 (0.7)
  Maximum Projection of Labia Majora Day 180 | 1.3 (0.3) | 0.9 (0.3)
  Arch of Labia Minora Day 180 | 8.7 (1.8) | 9.5 (1.0)
  Arch of Labia Majora Day 180 | 10.8 (1.5) | 10.5 (0.9)

3. Secondary Outcome: Analysis of Labia Protrusion (Distance of the Lateral Edge of the Labia Minora From That of the Labia Majora Rather Than the Introitus) at Baseline, D30, D90, and D180.
Description: MOTAKEF scale of labia protrusion, Type I-A: Less than 2cm, Type II-A: From 2cm to 4cm, Type II-C: From 2cm to 4cm, Type II-AI: From 4cm to 6 cm, Type VI-A: Greater than 6 cm. The greater the class the greater area of protrusion of labia minora past the labia majora. An "A" is added for asymmetry and a "C" for involvement of the clitoral hood.
Time Frame: Day 30, Day 90, Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Procedure with the Renuvion APR System in the labia (APR-15-TP) | Procedure with the Renuvion APR System in the labia (Micro)
Number analyzed (Participants) | 7 | 3
Participants
  Baseline: Type I-A: Less than 2cm | 0 | 0
  Baseline: Type II-A: From 2cm to 4cm | 6 | 3
  Baseline: Type II-C: From 2cm to 4cm | 1 | 0
  Baseline: Type II-AI: From 4cm to 6 cm | 0 | 0
  Baseline: Type VI-A: Greater than 6 cm | 0 | 0
  Day 30: Type I-A: Less than 2cm | 3 | 2
  Day 30: Type II-A: From 2cm to 4cm | 4 | 1
  Day 30: Type II-C: From 2cm to 4cm | 0 | 0
  Day 30: Type II-AI: From 4cm to 6 cm | 0 | 0
  Day 30: Type VI-A: Greater than 6 cm | 0 | 0
  Day 90: Type I-A: Less than 2cm | 3 | 2
  Day 90: Type II-A: From 2cm to 4cm | 4 | 1
  Day 90: Type II-C: From 2cm to 4cm | 0 | 0
  Day 90: Type II-AI: From 4cm to 6 cm | 0 | 0
  Day 90: Type VI-A: Greater than 6 cm | 0 | 0
  Day 180: Type I-A: Less than 2cm | 5 | 2
  Day 180: Type II-A: From 2cm to 4cm | 2 | 1
  Day 180: Type II-C: From 2cm to 4cm | 0 | 0
  Day 180: Type II-AI: From 4cm to 6 cm | 0 | 0
  Day 180: Type VI-A: Greater than 6 cm | 0 | 0

4. Secondary Outcome: Analysis of Hypertrophy of the Labia Minora (Hipertrofia de Ninfas) at Baseline, D30, D90, and D180
Description: Hipertrofia de Ninfas scale of hypertrophy; Type I (Less than 2cm), Type II (2-4cm), Type III (4-6cm), Type IV (<6cm). The lower the type the better the outcome.
Time Frame: Day 30, Day 90, Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Procedure with the Renuvion APR System in the labia (APR-15-TP) | Procedure with the Renuvion APR System in the labia (Micro)
Number analyzed (Participants) | 7 | 3
Participants
  Baseline: Type I: Less than 2cm | 0 | 0
  Baseline: Type II: From 2cm to 4cm | 7 | 3
  Baseline: Type III: From 4cm to 6 cm | 0 | 0
  Baseline: Type VI: Greater than 6 cm | 0 | 0
  Day 30: Type I: Less than 2cm | 3 | 2
  Day 30: Type II: From 2cm to 4cm | 4 | 1
  Day 30: Type III: From 4cm to 6 cm | 0 | 0
  Day 30: Type VI: Greater than 6 cm | 0 | 0
  Day 90: Type I: Less than 2cm | 2 | 2
  Day 90: Type II: From 2cm to 4cm | 5 | 1
  Day 90: Type III: From 4cm to 6 cm | 0 | 0
  Day 90: Type VI: Greater than 6 cm | 0 | 0
  Day 180: Type I: Less than 2cm | 5 | 2
  Day 180: Type II: From 2cm to 4cm | 2 | 1
  Day 180: Type III: From 4cm to 6 cm | 0 | 0
  Day 180: Type VI: Greater than 6 cm | 0 | 0

5. Secondary Outcome: The Subject Will Complete a Patient Satisfaction Questionnaire (PSQ) at the Day 180 Follow-up Visit.
Description: The subjects completed a Patient Satisfaction Questionnaire (PSQ) at the Day 180 follow-up visit. The subject completed this assessment while referring to baseline photos, current photos, and a hand mirror.
Time Frame: Day 180
Measure: Number; unit: participants
Arm/Group | Procedure with the Renuvion APR System in the labia (APR-15-TP) | Procedure with the Renuvion APR System in the labia (Micro)
Number analyzed (Participants) | 7 | 3
participants
  Do you notice improvement in how your labia look? : Yes | 7 | 3
  Characterize Satisfaction With Procedure - Satisfied (Very, Satisfied, or Slightly) | 6 | 3
  Recommend Procedure To Friends and Family Members - Yes | 6 | 3
  Improvement noticed - Closer together | 1 | 1
  Improvement noticed - Improvement in loose skin | 4 | 3
  Improvement noticed - Less sagging skin | 3 | 3
  Improvement noticed - Majora seem smaller-Right Minora seems same or only slight improvement | 1 | 1
  Improvement noticed - Smoother skin texture | 2 | 1

6. Secondary Outcome: During Study Treatment, the Subject's Pain Levels Will be Monitored Using the 11-point Numeric Rating Scale (NRS).
Description: During study treatment, the subject's pain levels were monitored using the 11-point Numeric Rating Scale (NRS). The average pain score for the entire region treated was recorded. Pain scores will be recorded at all follow-up visits. NRS 11-point Scale where 0 is no pain and 10 is most pain.
Time Frame: Post-Treatment, Day 1, Day 14, Day 30, Day 90, Day 180
Measure: Median (Standard Deviation); unit: Score on a Scale
Arm/Group | Procedure with the Renuvion APR System in the labia (APR-15-TP) | Procedure with the Renuvion APR System in the labia (Micro)
Number analyzed (Participants) | 7 | 3
Score on a Scale
  Baseline | 0.3 (0.8) | 0.0 (0.0)
  Day 1 | 4.1 (2.5) | 2.3 (2.1)
  Day 14 | 3.7 (3.4) | 4.0 (1.0)
  Day 30 | 1.6 (1.8) | 2.0 (0.0)
  Day 90 | 0.1 (0.4) | 0.0 (0.0)
  Day 180 | 0.0 (0.0) | 0.0 (0.0)

7. Secondary Outcome: The Principal Investigator, Sub-investigator or Qualified Clinician Delegated by the Principal Investigator, Will Complete a Bilateral Global Aesthetic Improvement Scale (GAIS) Assessing Overall Aesthetic Improvement in the Treatment Area.
Description: The Principal Investigator, sub-investigator or qualified clinician delegated by the principal investigator, completed a bilateral GAIS assessing overall aesthetic improvement in the treatment area at Day 30, Day 90, and Day 180 post-treatment.
  Global Aesthetic Improvement Scale: Very Much Improved, Much Improved, Improved, No Change, Worse, Much Worse, Very Much Worse
Time Frame: Day 30, Day 90, Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Procedure with the Renuvion APR System in the labia (APR-15-TP) | Procedure with the Renuvion APR System in the labia (Micro)
Number analyzed (Participants) | 7 | 3
Participants
  Day 30: Worse | 0 | 0
  Day 30: No Change | 2 | 0
  Day 30: Improved, Much Improved, Very Much Improved | 5 | 3
  Day 90: Worse | 0 | 0
  Day 90: No Change | 1 | 0
  Day 90: Improved, Much Improved, Very Much Improved | 6 | 3
  Day 180: Worse | 0 | 0
  Day 180: No Change | 0 | 0
  Day 180: Improved, Much Improved, Very Much Improved | 7 | 3

8. Secondary Outcome: The Subject Will Complete a GAIS Assessing Overall Aesthetic Improvement in the Treatment Area.
Description: The subject completed a GAIS assessing overall aesthetic improvement in the treatment area at Day 30, Day 90, and Day 180 post-treatment.
  Global Aesthetic Improvement Scale: Very Much Improved, Much Improved, Improved, No Change, Worse, Much Worse, Very Much Worse
Time Frame: Day 30, Day 90, Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Procedure with the Renuvion APR System in the labia (APR-15-TP) | Procedure with the Renuvion APR System in the labia (Micro)
Number analyzed (Participants) | 7 | 3
Participants
  Day 30: Worse | 0 | 0
  Day 30: No Change | 2 | 1
  Day 30: Improved, Much Improved, Very Much Improved | 5 | 2
  Day 90: Worse | 0 | 0
  Day 90: No Change | 0 | 1
  Day 90: Improved, Much Improved, Very Much Improved | 7 | 2
  Day 180: Worse | 0 | 0
  Day 180: No Change | 1 | 0
  Day 180: Improved, Much Improved, Very Much Improved | 6 | 3

9. Secondary Outcome: The Subject Will Complete a Female Sexual Function Index (FSFI) to Assess the Sexual Function to Evaluate the Impact of Treatment to the Labia.
Description: Female Sexual Function Index (FSFI) evaluation which measures desire, arousal, lubrication, orgasm, satisfaction, and pain, was administered at baseline, Day 90, and Day 180; 5 Answers available per question. The individual domain scores and full-scale score of the FSFI are derived by the computational formula. Response options for questions were: 0=no sexual activity, 5=almost always or always, 4=most times (more than half the time), 3=sometimes (about half the time), 2=a few times (less than half the time), 1=almost never or never. Individual domain scores are obtained by adding the scores of the individual items that comprise the domain and multiplying the sum by the specified domain factor. The full-scale score is obtained by adding the six domain scores with potential ranges from 2 to 36.
Time Frame: Baseline, Day 90, Day 180
Measure: Median (Standard Deviation); unit: Score on FSFI Scale (Range 2 - 36)
Arm/Group | Procedure with the Renuvion APR System in the labia (APR-15-TP) | Procedure with the Renuvion APR System in the labia (Micro)
Number analyzed (Participants) | 7 | 3
Score on FSFI Scale (Range 2 - 36)
  FSFI Baseline | 24.45 (1.1) | 25.17 (0.5)
  FSFI Day 90 | 24.45 (1.1) | 27.89 (1.3)
  FSFI Day 180 | 29.49 (0.8) | 26.51 (1.6)

10. Secondary Outcome: The Subject Will Complete a Genital Appearance Satisfaction (GAS) at Baseline, 90, and 180-day Follow-up Visits
Description: The Genital Appearance Satisfaction (GAS) scale was used to assess the satisfaction of subjects with their genital appearance following treatment to the labia at baseline, Day 90, and Day 180. The higher the GAS score reveals the greater dissatisfaction. Response options for each section of questions were Never (score 3), Sometimes (score 2), Often (score 1), Always (score 0). Question response values were added together for a final score for each participant. The best response would be 0 (no dissatisfaction). The worse response would be 30 (dissatisfaction across all questions).
Time Frame: Baseline, Day 90, Day 180
Measure: Mean (Standard Deviation); unit: Score on GAS Scale (0 -30 Range)
Arm/Group | Procedure with the Renuvion APR System in the labia (APR-15-TP) | Procedure with the Renuvion APR System in the labia (Micro)
Number analyzed (Participants) | 7 | 3
Score on GAS Scale (0 -30 Range)
  Genital Appearance Satisfaction Baseline | 18.57 (0.6) | 22.33 (0.5)
  Genital Appearance Satisfaction Day 90 | 9.14 (0.5) | 12.33 (0.4)
  Genital Appearance Satisfaction Day 180 | 9.86 (0.6) | 10.67 (0.5)

11. Secondary Outcome: Analysis of Days Until Subject Was Comfortable Returning to Sex.
Description: Subjects report the number of days until they feel comfortable returning to sex.
Time Frame: Post-Treatment, Day 1, Day 14, Day 30, Day 90, Day 180
Measure: Median (Standard Deviation); unit: Days
Arm/Group | Procedure with the Renuvion APR System in the labia (APR-15-TP) | Procedure with the Renuvion APR System in the labia (Micro)
Number analyzed (Participants) | 7 | 3
Days | 35.7 (26) | 21.7 (8.02)

ADVERSE EVENTS:
Time Frame: 180 Days
Description: An expected treatment effect (ETE) was defined as any typical treatment side-effect of Renuvion APR System of mild to moderate severity and lasting up to a typical maximum duration. An adverse event (AE) was defined as any new medical problem, or exacerbation of an existing problem, experienced by a subject while enrolled in the study, whether or not it is considered device-related by the investigator.
Arm/Group | Procedure With the Renuvion APR System in the Labia (APR-15-TP) | Procedure With the Renuvion APR System in the Labia (Micro)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/3
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Procedure With the Renuvion APR System in the Labia (APR-15-TP) (N=7) | Procedure With the Renuvion APR System in the Labia (Micro) (N=3)
Crepitus (ETE) (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (3)
Bruise (ETE) (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Edema (ETE) (Surgical and medical procedures) | 7 (7) | 3 (3)
Hypoesthesia/Numbness (ETE) (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (3)
Pain/Tenderness (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Pruritus/Itching (ETE) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Wound (Surgical and medical procedures) | 3 (3) | 0 (0)
Hematoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Hematoma

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the Principal Investigator and the Sponsor that restricts the PI's rights to discuss or publish trial results after the trial is completed. The data produced by this sponsored study is the sole property of Sponsor. Sponsor must be provided with the opportunity to review all Investigator-prepared abstracts, publications, or presentations for a period of thirty (30) days for presentational materials and abstracts and forty-five (45) days for manuscripts.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT05323630/Prot_SAP_000.pdf